CLINICAL TRIAL: NCT04145986
Title: Evaluation of Prognostic Monitoring for Young Breast Cancer Patients Via Analysis of Immunoinflammation-related Protein Complexes in Blood
Brief Title: Evaluation of Prognostic Monitoring for Young Breast Cancer Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Principal Investigator, Na Shi, Principal Investigator, Peking Union Medical College Hospital
Other Study IDs: PUMCH-BC503
Record Dates: First submitted 2019-10-29; First posted 2019-10-31 (Actual); Last update posted 2019-11-18 (Actual); Status verified 2019-11

CONDITIONS: Breast Cancer Female

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — 1 mL of blood
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- young ladies: Young ladies≤ 35 years old.

SUMMARY:
The relationship between immune inflammation-related protein complexes in blood and recurrence or metastasis of breast cancer with completed standard treatment for young ladies will be studied.

DETAILED DESCRIPTION:
200 patients younger than 35 with breast cancer will be followed up. Peripheral venous blood was collected every 3 to 6 months. Change regularity of breast cancer-specific immune inflammation-related protein complexes in blood at different follow-up time points will be studied. The relationship between disease specific protein complexes and pathological state of patients will be analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Female
* invasive breast cancer patients confirmed by postoperative pathology after surgery for breast lump
* Breast cancer-related chemotherapy and radiotherapy completed
* Young ladies with ages equal 35 or below

Exclusion Criteria:

* Male
* Aged above 35
* Breast Carcinoma in situ
* Women in pregnancy or breastfeeding
* Suffering from other malignant tumors
* Non-compliant patient

Max Age: 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Gender Based: Yes — The participant eligibility is based on the physiological sex.
Study Population: Breast cancer patients with ages equal 35 or below.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2019-04-25 (Actual); Primary Completion 2020-03 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
immune inflammation-related protein complexes | 2 years
  The change of immune inflammation-related protein complexes which is measured by gel permeation chromatography.
blood markers | 2 years
  The expression of CA153, CEA, CA125 in the blood of the patients, which are measured by electro-chemiluminescence immunoassay.

CONTACTS AND LOCATIONS:
Overall Officials: Shi Na, Principal Investigator — Peking Union Medical College Hospital
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China